CLINICAL TRIAL: NCT05777096
Title: Prevalence of Non-traumatic Musculoskeletal Disorders in the French Paragliding Pilots Population
Acronym: EPPPAF
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A00131-44
Record Dates: First submitted 2023-03-07; First posted 2023-03-21 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Prevalence; Musculoskeletal Disorders
Keywords: paragliding; musculoskeletal Diseases; non-traumatic pathology; Standardised Nordic Questionnaire; overuse injury
MeSH Terms: conditions — Musculoskeletal Diseases; Cumulative Trauma Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- registered: Paragliding pilots over the age of 18. Registered at the "Fédération Française de Vol Libre" (FFVL) in the year 2022 and/or 2023 Paragliding in the year 2022 and/or 2023
  Interventions: Diagnostic Test: Standardised Nordic questionnaires

INTERVENTIONS:
Diagnostic Test: Standardised Nordic questionnaires — participants will complete the SNQ online. Estimated time of participation per person: 15 minutes to fill in the questionnaires

SUMMARY:
The main objective is to determine the prevalence of non-traumatic pathologies in the paragliding population using the Nordic type questionnaire.

The paragliding pilots population frequently evoque pathologies, discomfort, or pain in the course of their practice. Said pain and discomfort, though unerelated any form of accident, seem to have an impact on the pilots' flying and their participation in daily life.

However, no epidemiological data are available in the literature. Investigators hypothesize the existence of non-traumatic disorders and it seems interesting to quantify the extent of the phenomenon. The results of this study might encourage the proposition of preventive measures in order to minimize a potential risk factor for paragliding accidents, and participation restrictions.

DETAILED DESCRIPTION:
In this cross-sectional descriptive epidemiological survey, investigators wish to quantify epidemiological parameters such as the prevalence of pathologies and their consequences in the activities of daily life.

For this purpose, an email containing the link to answer the online questionnaire will be sent to all the licensees.

The link of the questionnaire will be sent directly to all clubs in each league.

The main objective is to calculate the prevalence with descriptive statistics. The primary outcome is the prevalence of non-traumatic pathology in paragliding pilots that had registered to the French Paragliding federation (FFVL) in 2022.

The prevalence will be infered from the IRSST Standardised Nordic Questionnaire with the following formula : Prevalence = (FS4+FS6=yes and FS2=no ) divided by the total number of respondents.

FS4 item "Yes" = pain in the last 12 months FS6 item "Yes" = activity limitations) FS2 item "No" = Non-traumatic disorders

This corresponds to having felt pain in the body region indicated, at least once during the last 12 months, as well as a restriction of participation following this pain, but without having suffered trauma in the area.

For the secondary outcomes will aim at exploring several hypotheses related to personal and environmental factors that could be correlated to the incidence of the nontraumatic disorders. They will be calculated with bivariate descriptive statistics using the Pvalue.io software.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* Registered with the FFVL for the year 2022 and/or 2023
* Paragliding in the year 2022 and/or 2023

Exclusion Criteria:

* Adults not able to express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 26000 people will be surveyed via the internet link. In 2021, according to the federal statistics of the FFVL accessible on the intranet of the FFVL, the number of practicing paraglider with a license was about 26000.
Sampling Method: Non-Probability Sample
Enrollment: 2475 (Actual)
Dates: Start 2023-03-12 (Actual); Primary Completion 2023-06-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of non-traumatic pathologies in the paragliding pilot population | Cross sectional study. Each participant is evaluated for 15 minutes (estimated time of completion of the questionnaire)
  The prevalence will be calculated using the IRSST's Standardised Nordic Questionnaire.
  Prevalence = (FS4+FS6=yes and FS2=no ) on total number of respondents. This prevalence will be calculated on the Population Health, with the FS4 and FS6 items. And to be more specific about atraumatic pathologies, it is necessary to have answered "no" to the FS2 item. This corresponds to having felt pain in the body region indicated, at least once during the last 12 months, as well as a restriction of participation following this pain, but without having undergone trauma in the area concerned.

SECONDARY OUTCOMES:
Correlations between prevalence, a body area, restriction of participation in paragliding and individual characteristics of participants | Cross sectional study. Each participant is evaluated for 15 minutes (estimated time of completion of the questionnaire)
  Correlation analysis (univariate and bivariate) between responses to different questions to test for a potential association between variables
Paragliders' beliefs about the origin of their pain. | Cross sectional study. Each participant is evaluated for 15 minutes (estimated time of completion of the questionnaire)
  Number of respondents with musculoskeletal disorder (FS9=yes)/total number of positive cases ((FS4+FS6=yes and FS2=no)
Prevalence of injuries sustained during a paragliding accident | Cross sectional study. Each participant is evaluated for 15 minutes (estimated time of completion of the questionnaire)
  Number of respondents with musculoskeletal disorder due to accident/total number of pain positive cases and participation restriction ((FS4+FS6=yes and FS2.3=yes)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas LATHIERE, Principal Investigator — Département de kinésithérapie, 175 avenue centrale 38400 Saint Martin d'Hères
Locations (1):
- Grenoble Alpes University - Faculty of Medecine - Departement of Physiotherapy, Saint-Martin-d'Hères, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuorinka I, Jonsson B, Kilbom A, Vinterberg H, Biering-Sorensen F, Andersson G, Jorgensen K. Standardised Nordic questionnaires for the analysis of musculoskeletal symptoms. Appl Ergon. 1987 Sep;18(3):233-7. doi: 10.1016/0003-6870(87)90010-x. PMID 15676628
- [Background] desLibris, L'enquête québécoise sur la santé de la population 2008, Canadian Electronic Library. Canada. Retrieved from https://canadacommons.ca/artifacts/1238967/lenquete-quebecoise-sur-la-sante-de-la-population-2008/1792039/ on 05 Mar 2023. CID: 20.500.12592/rvf74g.
- [Background] Alexis Descatha, Yves Roquelaure, Agnès Aublet-Cuvelier, Catherine Ha, Annie Touranchet, et al.. Validité du questionnaire de type "Nordique" dans la surveillance des pathologies d'hypersollicitation du membre supérieur. Documents pour le Médecin du Travail, 2007, pp.509-517. ffinserm-00232629
- See also: Sample size for a prevalence survey, with finite population correction — http://sampsize.sourceforge.net/iface/index.html